CLINICAL TRIAL: NCT06732583
Title: A Phase I Randomized, Double-blind, Placebo-controlled and Dose Escalation Study to Evaluate the Safety and Immunogenicity of a Viral Vector-based Tuberculosis (TB) Vaccine Ad5-105K Against TB Disease in Adults Aged 18 to 49 Years
Brief Title: A Study to Evaluate the Safety and Immunogenicity of Ad5-105K in Adults Aged 18 to 49 Years
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Collaborators: PT Etana Biotechnologies Indonesia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTP-ADTB-001
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Tuberculosis
Keywords: Vaccine; Ad5-105K; Immunogenicity; Safety; 18-49 years; TB
MeSH Terms: conditions — Tuberculosis | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental vaccine group, Low dose (Experimental): 1 doses of Ad5-105K vaccine (0.1ml) on Day 0
  Interventions: Biological: Tuberculosis (TB) vaccine (Ad5-105K)
- Placebo Group, Low dose (Placebo Comparator): 1 doses of placebo (0.1ml) on Day 0
  Interventions: Biological: Placebo
- Experimental vaccine group, High dose (Active Comparator): 1 doses of Ad5-105K vaccine (0.2ml) on Day 0
  Interventions: Biological: Ad5-105K
- Placebo Group, High dose (Placebo Comparator): 1 doses of placebo (0.2ml) on Day 0
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Tuberculosis (TB) vaccine (Ad5-105K) — 1 doses of Ad5-105K vaccine (1 x 10^8 vp)) on Day 0, Nebulized Inhalation (IH) through mouth
  Arms: Experimental vaccine group, Low dose
Biological: Placebo — 1 doses of placebo on Day 0, IH
  Arms: Placebo Group, Low dose
Biological: Ad5-105K — 1 doses of Ad5-105K vaccine (2 x 10^8 vp)) on Day 0, IH
  Arms: Experimental vaccine group, High dose
Biological: Placebo — 1 doses of placebo on Day 0, IH
  Arms: Placebo Group, High dose

SUMMARY:
This is a randomized, observer-blind, positive-controlled study. There will be 2 treatment groups (Group A and B). In each treatment group, 18 participants will be randomly assigned to receive either the investigational vaccine (Dose A or Dose B of Ad5-105K) or a placebo in a ratio of 2:1. The distribution of participant's gender and age should be balanced in each group.

ELIGIBILITY:
Inclusion Criteria:

* Participants who, in the opinion of the investigator, are able and willing to comply with the requirements of the protocol (e.g., completion of diary cards, returning for follow-up visits).
* Healthy male or female participants aged 18 to 49 years, at the time of obtaining informed consent.
* Written (or thumb printed and witnessed) informed consent obtained from the participant.
* Positive IGRA test with no history of TB disease or treatment.
* Female participants of childbearing potential must have a negative urine pregnancy test at screening and on the day of vaccination. Male and female participants of childbearing potential must agree to use adequate contraception for the entire duration of their participation in the study.
* History of BCG vaccination.

Exclusion Criteria:

* Current TB disease, or a history of TB disease and/or treatment for TB (including Tuberculosis Preventive Therapy (TPT)).
* Known history of close or household contact with active TB patient.
* Axillary temperature ≥37.5°C.
* Presence of congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.
* Lactating women.
* Individuals who smoke more than 10 cigarettes per day within the last 3 months and/or more than 2 cigars per day, and/or vapers who use more than 5 ml of e-liquid daily.
* Individuals with positive HIV, HBV, HCV, or TP (Treponema pallidum) test.
* History of immunosuppressive treatment, cytotoxic treatment, or glucocorticoid treatment, etc. (excluding local treatments, surface treatments for acute non-concurrent dermatitis or spray treatment for allergic rhinitis) in the past 6 months (internal time <6 months).
* History of, or plans to use, blood/plasma products or immunoglobulins within 60 days prior to study vaccination or at any time during the study period.
* Uncontrolled severe hypertension (at the time of field measurement: systolic blood pressure ≥160 mmHg and diastolic blood pressure ≥100 mmHg).
* Suffering from a serious chronic disease or a condition that is in a progressive stage and cannot be adequately controlled (e.g., thyroid disease), or having known or suspected diseases that at investigators' discretion, may affect vaccination or immunogenicity test results (e.g., diagnosed with asthma within the last 20 years, severe respiratory disease, acute infection or active chronic disease, severe cardiovascular disease, severe liver or kidney disease, malignancy, severe infectious or allergic skin disease).
* History of serious adverse reactions associated with the adenovirus vector-based vaccine and/or history of severe allergic reactions (e.g., systemic allergic reactions) to any component of the study vaccine.
* Immunocompromised individuals with known or suspected immunodeficiency as determined by medical history and/or physical examination (e.g., HIV infection, or a history of pancreatic, liver, spleen, kidney disease, or a history of organ resection).
* Bleeding constitution or condition associated with prolonged bleeding for which IM injection is contraindicated, in the opinion of the investigator.
* History of administration of any vaccine within the past three months.
* History of receiving experimental Mycobacterium tuberculosis (Mtb) vaccines or participation in other interventional studies within 28 days prior to screening and/or during study participation.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Occurrence of solicited adverse events (AEs) | Within 7 days after vaccination

SECONDARY OUTCOMES:
Occurrence of solicited AEs | Within 30 mins after vaccination
Occurrence of unsolicited AEs | Within 28 days after vaccination
Occurrence of serious adverse events (SAEs) and adverse events of special interest (AESI) | Through study completion, an average of 6 months
Occurrence of abnormal hematology and chemistry laboratory assessments | On Day 3 after vaccination
Geometric mean titer (GMT) of anti-TB75K and anti-Ag85A IgG antibodies before vaccination | On Day 14 and Day 28 post-vaccination
Expression level of IFN-γ, TNF-α, IL-2, and IL-17 in 105K specific CD4+/CD8+ T cells evaluated by ICS | Before vaccination and on Day 14 and Day 28 post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Erlina Burhan, Principal Investigator — Respiratory Programmatic Implementation and Research Institute & RSUP Persahabatan
Locations (1):
- Rumah Sakit Islam Jakarta Cempaka Putih, Jakarta, Indonesia